CLINICAL TRIAL: NCT05465109
Title: Designing and Evaluating a Comprehensive Support Program for Families Caring for Relatives Living With TBI-AD/ADRD
Brief Title: Traumatic Brain Injury and Alzheimer's Disease/Related Dementias Caregiver Support Intervention
Acronym: TACSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); Mayo Clinic (Other); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00014886; CDMRP-AZ200106 (Other: CDMRP)
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Caregiver Burden; Caregiver Stress Syndrome; Caregiver Burnout
Keywords: Caregiver; Traumatic brain injury; Alzheimer's; Dementia
MeSH Terms: conditions — Caregiver Burden; Brain Injuries, Traumatic; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACSI (Experimental)
  Interventions: Other: TBI-AD/ADRD Caregiver Support Intervention (TACSI)
- Usual care control group (No Intervention): The usual care control group would have continued receipt of standard services at either the Mayo Clinic or the MVAHCS. In addition, staff will offer participants the opportunity to request supportive/educational resources as needed after randomization.

INTERVENTIONS:
Other: TBI-AD/ADRD Caregiver Support Intervention (TACSI) — The TBI-AD/ADRD Caregiver Support Intervention (TACSI) incorporates psychosocial and psychoeducational approaches with the objective of: a) identifying stressors associated with caregiving for family members who have the dual diagnosis of traumatic brain injury and dementia; and b) supporting caregivers in developing more effective coping and communication strategies as well as enhanced caregiving self-efficacy. This intervention offers individual and family coaching and knowledge and skills to help manage stress and reduce caregiver burden.
  Arms: TACSI

SUMMARY:
The TBI-AD/ADRD Caregiver Support Intervention (TACSI) incorporates psychosocial and psychoeducational approaches with the objective of: a) identifying stressors associated with caregiving for family members who have the dual diagnosis of traumatic brain injury and dementia; and b) supporting caregivers in developing more effective coping and communication strategies as well as enhanced caregiving self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* the care recipient has a physician diagnosis of TBI and AD/ADRD (i.e., those with a diagnosis of both TBI and progressive cognitive decline)
* the caregiver self-identifies as someone who provides the most help/is most responsible for the person with TBI-AD/ADRD because of their cognitive impairments (or shares the role equally with another caregiver)
* the caregiver indicates a willingness to participate in the TACSI evaluation
* the caregiver is English speaking
* the caregiver is 21 years of age or older
* the caregiver is not currently participating in any other type of service that provides one-to-one psychosocial consultation or caregiver coaching (peer mentorship/support group participation/general counseling not specific to caregiving is not a deterrent to enrollment) at the discretion of the UMN research team
* the caregiver resides in the US.

Exclusion Criteria:

* caregivers who have a new or worsening mental health condition and are not receiving ongoing treatment. When applicable, if caregivers have not remained on a stable psychotropic medications dosage, such as antidepressants, anxiolytics or anti-psychotics, for the prior three months they will be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-28 (Actual); Study Completion 2025-06-28 (Actual)

PRIMARY OUTCOMES:
Caregiver primary subjective stress- Phase 1 | change in score from baseline to 3 months
  Change in score from baseline to Module 6
Caregiver primary subjective stress- Phase 2, 3mo | change in score from baseline to 3 months
  Change in score from baseline to Module 6
Caregiver primary subjective stress- Phase 2, 6mo | change in score from baseline to 6 months
  Change in score from baseline to Module 6

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT05465109/ICF_001.pdf